CLINICAL TRIAL: NCT00418262
Title: An Open-label Study of the Long Term Tolerability and Safety of Atomoxetine in Treating the Inattention, Impulsivity and Hyperactivity in Children With Fetal-Alcohol Syndrome or Effects.
Brief Title: Open-Label Study of the Long Term Tolerability and Safety of Atomoxetine in Children With FASD and ADD/ADHD
Acronym: B4Z-US-050
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Mark L. Wolraich (Unknown)
Responsible Party: Principal Investigator, Laura J McGuinn, MD, Principal Investigator, University of Oklahoma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2112
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Fetal Alcohol Syndrome; Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: fetal alcohol syndrome; attention deficit disorder; attention deficit disorder with hyperactivity; ADD; FAS; FASD; ADHD
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atomoxetine HCL (Strattera) (Experimental): Teatment of children with fetal alcohol syndrome and ADHD with Atomoxetine HCL (Strattera)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Titrating with oral administration of 0.25 mg/kg, 0.50 mg/kg, 1.0 mg/kg, or 1.4 mg/kg once each morning with food.
  Other Names: Brand Name: Strattera, Serial Number: 76306506, ACT

SUMMARY:
Determine if atomoxetine is safe and well tolerated by children with fetal alcohol syndrome.

DETAILED DESCRIPTION:
Abnormalities of attention, function, and activity level in children exposed to alcohol in utero share similarities and differences to children who do not have alcohol exposure. Previous psychological studies have examined either core attention deficit hyperactivity (ADHD) symptoms of hyperactivity, inattention, and impulsivity or hypothesized neuropsychological differences in children with fetal alcohol syndrome (FAS) and ADHD. Atomoxetine Hydrochloride is a non-stimulant medication used to treat ADHD. This study will determine if atomoxetine HCL significantly reduces symptoms of ADD/ADHD in children with fetal alcohol exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been between the ages of 4 and 11 years at the time of entry into the double blind study.
* Patients must meet diagnostic criteria for FASD.
* Patient must, at entry into doubleblind study, have met DSM-IV criteria for ADHD, any subtype. And must have an ADHDRS-IV score of > or + 90% for age and gender on either subtest or total score for children above 5 years of age.
* Patients will continue atomoxetine/placebo until entry nto this study.
* History and physical exam must reveal no clinically significant abnormalities that would preclude safe participation in the study.
* Patients must be able to swallow capsules.
* Patients must be of a sufficient mental age (3 yrs) to participate in the study.
* Patients and parents must be able to communicate effectively with the investigator and coordinator and be judged reliable to keep appointments and participate in data collection.
* Teacher must agree to cooperate with the study.

Exclusion Criteria:

* Have received an investigational medication other than atomoxetine in the previous 30 days.
* Have significant current medical conditions that could be exacerbated or compromised by atomoxetine.
* Have used MAOIs within one month prior to visit 1.
* Patients with hypertension.
* Patients with a previous diagnosis of bipolar disorder, psychosis, or autism spectrum disorder.
* Patients taking anticonvulsants for seizure control.
* Patients taking another psychotropic medication or health food supplements purported to have central nervous system activity within 5 half-lives of visit 1.
* Patients with Tourette Disorder or any other neurological condition that would interfere with their ability to receive treatment or comply with monitoring.
* Pubertal girls.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura J McGuinn, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- OU Child Study Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study the recruited 29 (21 male/8 female) children between 10/18/2006 and 9/21/2011. The children were recruited from a prior efficacy trial. Participants for the efficacy trial were drawn from physician referral resources, self-referral, and a pool of subjects identified for a study sponsored by the Center for Disease Control and Prevention.
Pre-assignment Details: Two recruits declined particicpation in this open-label study. Participants continued to take atomoxetine/placeblo (depending on prior RCT assignment) until entry into this open label study.
Groups:
- Atomoxetine HCL (Strattera): The subjects will receive atomoxetine at 0.5 mg/kg/day for the first week. The children will be seen weekly for assessment for 4 weeks, every month for two months, then every three months until the 12 month treatment period is complete. After one week of treatment response will be reassessed and the dose will be increased to 1.0 mg/kg/d unless there are excessive side effects. If there are mild side effects the dose will be held the same. If there are excessive side effects the dose will be split to 0.25 mg/kg-d BID. At visit 3 the dose will be increased to 1.0 or 1.4 mg/kg-d, depending on the previous dose, if there are not excessive side effects. This titration will occur at each visit.
Period: Visits 1 (Baseline) Thru 5
Arm/Group | Atomoxetine HCL (Strattera)
Started | 27
Completed | 25
Not Completed | 2
Period: Visits 5 Thru 8
Arm/Group | Atomoxetine HCL (Strattera)
Started | 25
Completed | 16
Not Completed | 9
Period: Visits 8 Thru 10
Arm/Group | Atomoxetine HCL (Strattera)
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine HCL (Strattera): The subjects will receive atomoxetine at 0.5 mg/kg/day for the first week. The children will be seen weekly for assessment for 4 weeks, every month for two months, then every three months until the 12 month treatment period is complete. After one week of treatment response will be reassessed and the dose will be increased to 1.0 mg/kg/d unless there are excessive side effects. If there are mild side effects the dose will be held the same. If there are excessive side effects the dose will be split to 0.25 mg/kg-d BID. At visit 3 the dose will be increased to 1.0 or 1.4 mg/kg-d, depending on the previous dose, if there are not excessive side effects. This "titration" will occur at each visit.
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.4 [4.3 to 12.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | NA — Not assessed
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Pittsburg Side-Effects Scale: Motor Tics
Description: Motor Tics
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: Children with FAS participating in the extend safety efficacy study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine HCL (Strattera): Treatment of children with fetal alcohol syndrome and ADHD with Atomoxetine HCL (Strattera)
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.15 (0.54)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.20 (0.50)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.31 (0.60)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.27 (0.47)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); Tested single-group change over time from baseline (visit 1) to the study endpoint (visit 10). The null hypothesis stated that there was no change in PSE ratings over time. Bayesian growth curve models were estimated using Markov Chain Monte Carlo techniques. Several linear and nonlinear trajectory models were compared on fit to data. Mean differences and confidence intervals were generated from the posterior-predictive distribution of the "best" fitting growth model; Test type: Superiority; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.21 to 0.30] — This is the (growth) model-estimated mean difference between visit 1 and visit 8. This estimate utilizes imputed values for missing observations
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.42 to 0.60] — This is the (growth) model-estimated mean difference between visit 1 and visit 10. This estimate utilizes imputed values for missing observations

2. Primary Outcome: Pittsburg Side-Effects Scale-Buccal, Lingual Movements
Description: Buccal, Lingual Movements
  Parent rating of none (0), mild (1), moderate (2) or severe (3) for each manifestation.
Time Frame: 12 months or study duration
Population: Attrition
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | .12 (.33)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.2 (0.50)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.44 (0.73)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.27 (0.47)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.11 to 0.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.23 to 0.77] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Pittsburg Side-Effects Scale: Movements, Picking/Chewing Skin or Fingers
Description: Movements, Picking/Chewing Skin or Fingers
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: 27 IN PCT and one subject did not enroll in the safety efficacy study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.42 (0.70)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.40 (0.58)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.62 (0.89)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.64 (1.03)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.17 to 0.36] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.17 to 0.36] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Pittsburg Side-Effects Scale: Worried/Anxious
Description: Worried/Anxious
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject from RCT did not enroll in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine HCL (Strattera): Visit 1
  One additional subject left the study
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.27 (0.45)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.24 (0.60)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.56 (0.63)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.45 (0.69)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.16 to 0.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.16 to 0.40] — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Pittsburg Side-Effects Scale: Dull/Tired/Listless
Description: Dull/Tired/Listless
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject from the RCT did not enter the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atomoxetine HCL (Strattera): One additional subject left the study
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.31 (0.62)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.36 (0.57)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.38 (0.62)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.36 (0.50)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.36 to 0.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.36 to 0.18] — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Pittsburg Side-Effects Scale: Headaches
Description: Headaches
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject from the RCT did not enter the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.23 (0.51)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.40 (0.82)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.31 (0.60)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.18 (0.40)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.20 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.20 to 0.35] — [estimate comment as in outcome 1, analysis 2]

7. Primary Outcome: Pittsburg Side-Effects Scale: Stomachaches
Description: Stomachaches
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject in the RCT did not enroll in the Open Label Study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.23 (0.51)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.36 (0.49)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.25 (0.58)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.45 (0.82)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.24 to 0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.49 to 0.49] — [estimate comment as in outcome 1, analysis 2]

8. Primary Outcome: Pittsburg Side-Effects Scale: Crabby/Irritable
Description: Crabby/Irritable
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One Subject in the RCT did not enroll in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.85 (0.88)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.68 (0.85)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 1.06 (0.85)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.73 (0.65)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.28 to 0.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.56 to 0.52] — [estimate comment as in outcome 1, analysis 2]

9. Primary Outcome: Pittsburg Side-Effects Scale: Tearful/Sad/Depressed
Description: Tearful/Sad/Depressed
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject in RCT did not participate in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.19 (0.40)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.24 (0.52)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.50 (0.63)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.27 (0.47)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.32 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Median Difference (Net) = -0.12, 95% CI 2-sided [-0.64 to 0.39] — [estimate comment as in outcome 1, analysis 2]

10. Primary Outcome: Pittsburg Side-Effects Scale: Socially Withdrawn
Description: Socially Withdrawn
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject in the RCT did not enroll in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.12 (0.43)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.16 (0.47)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.25 (0.58)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.09 (0.30)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.28 to 0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.57 to 0.47] — [estimate comment as in outcome 1, analysis 2]

11. Primary Outcome: Pittsburg Side-Effects Scale: Hallucinations
Description: Hallucinations
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject in the RCT did not enroll in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.04 (0.20)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.00 (0.00)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.12 (0.50)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.00 (0.00)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.21 to 0.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.21 to 0.32] — [estimate comment as in outcome 1, analysis 2]

12. Primary Outcome: Pittsburg Side-Effects Scale: Loss of Appetite
Description: Loss of Appetite
  Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation
Time Frame: 12 months or study duration
Population: One subject in the RCT did not enroll in the open label study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.46 (.65)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.56 (0.65)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.38 (0.50)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.45 (0.52)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.36 to 0.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.22, 95% CI 2-sided [-0.72 to 0.27] — [estimate comment as in outcome 1, analysis 2]

13. Primary Outcome: Pittsburg Side-Effects Scale: Trouble Sleeping
Description: Trouble Sleeping Parent rating of none (0), mild (1) , moderate (2) or severe (3) for each manifestation.
Time Frame: 12 months or study duration
Population: One subject participating in the RCT did not participate in the open label
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 0.35 (0.57)
  Visit 5: number analyzed (Participants) | 25
  Visit 5 | 0.64 (0.70)
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 0.53 (0.74)
  Visit 10: number analyzed (Participants) | 11
  Visit 10 | 0.40 (0.52)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.19 to 0.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.19 to 0.35] — [estimate comment as in outcome 1, analysis 2]

14. Secondary Outcome: Determine if Changes in Behavior Seen With Short-term (Eight Weeks) Treatment of Children Are Maintained Over a Twelve Month Period.
Description: Parent rate the frequency of 18 of their child's behaviors from not at all (0), just a little (1) , pretty much (2) to very much (3) for each behavior. The Item scores were summed to arrive at a total score which ranged from 0 to 54. The higher the score, the worse the behavior.
Time Frame: 12 months or study duration
Population: ADHD Parent Rating Scale
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
units on a scale
  Visit 1 | 37.35 [32.64 to 42.35]
  Visit 8: number analyzed (Participants) | 16
  Visit 8 | 27.87 [23.52 to 32.26]
  Visit 10 | 31.88 [24.94 to 38.63]
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -7.40, 95% CI 2-sided [-7.76 to -7.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = -2.44, 95% CI 2-sided [-3.03 to -1.90] — [estimate comment as in outcome 1, analysis 2]

15. Secondary Outcome: Compare Growth While on Atomoxetine With Growth Before Entry Into Study.
Description: Height measured in centimeters at the time of each visit as part of the vital signs.
Time Frame: 12 months or study duration
Population: Measurements of height were not consistently obtained on all subjects.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Atomoxetine HCL (Strattera): Teatment of children with fetal alcohol syndrome and ADHD with Atomoxetine HCL (Strattera)
  atomoxetine hydrochloride: Titrating with oral administration of 0.25 mg/kg, 0.50 mg/kg, 1.0 mg/kg, or 1.4 mg/kg once each morning with food.
Arm/Group | Atomoxetine HCL (Strattera)
Number analyzed (Participants) | 26
cm
  Visit 1: number analyzed (Participants) | 23
  Visit 1 | 121.67 (9.84)
  Visit 8: number analyzed (Participants) | 3
  Visit 8 | 123.27 (4.01)
  Visit 10: number analyzed (Participants) | 7
  Visit 10 | 132.13 (8.77)
Statistical Analysis 1: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.69 to 1.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Atomoxetine HCL (Strattera); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.69 to 1.38] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Ccause Mortality and Serious Adverse Events were monitored.
Groups:
- Atomoxetine HCL (Strattera): The subjects received 7 days of atomoxetine at 0.5 mg/kg/day. The children were seen weekly for assessment for 4 weeks then every two weeks until the eight week double blind period was completed. After each week of treatment, response was reassessed and the dose was increased to 1.0 then 1.4 mg/kg/d unless there were excessive side effects. The subjects were then invited to continue for 1 year to assess safety and efficacy
Arm/Group | Atomoxetine HCL (Strattera)
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 19/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine HCL (Strattera) (N=26)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (204) — Cough
Vomiting (Gastrointestinal disorders) | 8 (204) — Vomiting
Headache (Nervous system disorders) | 8 (204) — Headache
Stomachache (Gastrointestinal disorders) | 7 (204) — Stomachache
Sleepy or Sleep Trouble (Nervous system disorders) | 7 (204) — Sleepy or Sleep Trouble
Nasal Congestion or Rhinorrhea (General disorders) | 6 (204) — Nasal Congestion or Rhinorrhea
Irritability (Psychiatric disorders) | 4 (204) — Irritability
Enuresis (Renal and urinary disorders) | 4 (204) — Enuresis
Fever (General disorders) | 4 (204) — Fever
Upper Respiratory or Sinus Infection (Infections and infestations) | 4 (204) — Upper Respiratory or Sinus Infection
Dizziness (General disorders) | 3 (204) — Dizziness
Diarrhea (Gastrointestinal disorders) | 3 (204) — Diarrhea
Ear Infection (Ear and labyrinth disorders) | 3 (204) — Ear Infection
Skin Rash or Redness (Skin and subcutaneous tissue disorders) | 2 (204) — Skin Rash or Redness
Sore Throat (Infections and infestations) | 2 (204) — Sore Throat
Decreased Appetite (Gastrointestinal disorders) | 2 (204) — Decreased Appetite
Asthma or Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (204) — Asthma or Wheezing
Fatigue (General disorders) | 2 (204) — Fatigue
Sad and Angry or Mood Swings (Psychiatric disorders) | 2 (204) — Sad and Angry or Mood Swings

LIMITATIONS AND CAVEATS:
There were a limited number of subjects because of difficulties in recruiting children with FAS and ADHD within the age group studied. We were only able to obtain a small number of teacher rating scales.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No